CLINICAL TRIAL: NCT01957631
Title: Steroid Injections vs. Platelet Rich Plasma Injections in Patients With Plantar Fasciitis: A Comparison of Clinical and Ultrasound Findings
Brief Title: Comparing Steroid Injections and Platelet Rich Plasma Injections in the Treatment of Plantar Fasciitis
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: King Hamad University Hospital, Bahrain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AJB88AK
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Plantar Fasciitis
Keywords: Plantar Fasciitis; Steroid; Platelet rich plasma; Injection; Ultrasound
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Adrenal Cortex Hormones; Bupivacaine; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corticosteroid injection (Active Comparator): Corticosteroid injection
  Interventions: Drug: Corticosteroid injection (Bupivacaine and Depo Medrol)
- Platelet rich plasma injection (Experimental): Platelet rich plasma injection
  Interventions: Biological: Platelet rich plasma injection

INTERVENTIONS:
Drug: Corticosteroid injection (Bupivacaine and Depo Medrol) — The use of corticosteroid injections to treat heel pain has been a relatively common practice. They are mainly used in conjunction with other modes of conservative therapies. With a 10cc syringe, 3 mL of 0.5% Bupivacaine and 2 mL of 80mg Depo Medrol are injected into the medial calcaneal tubercle using an aseptic technique.
  Other Names: Bupivacaine, Depo Medrol
  Arms: Corticosteroid injection
Biological: Platelet rich plasma injection — 10-15cc of patient's blood is drawn and centrifuged in a Rotofix 32A at 1500 cycles/minute for 5 minutes to separate the platelets from the other components of blood. 4-6cc of concentrated platelets are then re-injected into the medial calcaneal tuberosity using an aseptic technique. Sterile techniques are very important in this procedure to decrease the risk of infection.
  Arms: Platelet rich plasma injection

SUMMARY:
In cases of Plantar Fasciitis not responding to conservative management, minimally invasive techniques may be used. These include platelet rich plasma injections and corticosteroid injections. Corticosteroids have long been used for symptomatic relief. However there are growth factors present in PRP injections that contribute to the healing of the pathology, and not just symptom control.

A single blind, prospective, randomized, comparative, control study will be performed. The study population consists of a total of 80 participants. They will be randomly assigned to receive either a corticosteroid injection, or a platelet rich plasma injection. Data will be collected through questionnaires and ultrasound findings. Patients will have a follow up at 3, 6, 12, and 24 weeks after they receive their injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18+
* Patients with Plantar Fasciitis for at least 6 months which has not responded to 6 weeks of conservative therapy
* Patients with a visual analogue score (VAS) of more than 5 in the morning
* Patients must be able to understand the informed consent and have the ability to follow up.

Exclusion Criteria:

* Patients who have had repeated corticosteroid injections within the past 3 months, or have taken a non-steroid anti inflammatory drug during the 1 week prior to receiving an intervention
* BMI > 40
* Patients with a previous foot deformity
* Patients who have had previous foot surgery
* History of anemia (Hb < 7)
* Confirmed diagnosis of neuropathy
* Patients who have the inability to follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 6 months
  Pain will be measured using the visual analogue score (VAS). The score is a 10cm line, where each centimeter is marked between 0-10. Patients will mark the number that corresponds to their pain, where zero is no pain and 10 being the most severe pain.
  Every patient must at least have a pre and post intervention score recorded. Subsequent follow-ups will also require patients to fill out a VAS score. A 30% reduction between baseline and endpoint score over a period of 6 months, without the use of analgesia beyond what is allowed according to protocol, use of adjunctive conservative therapy (excluding physiotherapy), or the patient seeking alternative therapy, will deem the treatment successful. The reduction is calculated by subtracting the baseline value from the endpoint value. The percent change is determined by multiplying the reduction by 100 and dividing by 10.

SECONDARY OUTCOMES:
Ultrasound findings | 3 months
  All patients will have an ultrasound pre and three and six months post intervention. The thickness of the plantar fascia will be measured.
  Any decrease in the thickness will be taken into account and contributed to a successful intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ahsan J Butt, Principal Investigator — King Hamad University Hospital, Bahrain; Aamina M Khan, Principal Investigator — King Hamad University Hospital, Bahrain
Locations (1):
- King Hamad University Hospital, Al Muharraq, Bahrain